CLINICAL TRIAL: NCT01840709
Title: Effectiveness Study of Brief Group Psychoanalytic Psychotherapy (BGPP) to Improve Quality of Life in Patients With Systemic Lupus Erythematosus.
Brief Title: Effectiveness Study of Psychotherapy in Systemic Lupus Erythematosus
Acronym: PSYCHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Emilia Inoue Sato, MD, PhD - Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UNIFESP.PSYCHO
Record Dates: First submitted 2012-10-31; First posted 2013-04-26 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Psychotherapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychotherapy treatment (Experimental): The experimental group will be treated with Psychoanalytic brief group psychotherapy once a week for 20 consecutive weeks.
  Interventions: Behavioral: Psychotherapy
- control group (No Intervention): the patients in this group will be just assessed with the same questionnaires at baseline and after 20 weeks, without psychotherapy.

INTERVENTIONS:
Behavioral: Psychotherapy — Psychoanalytic brief group psychotherapy once a week for 20 consecutive weeks
  Arms: Psychotherapy treatment

SUMMARY:
Psychosomatic is a new approach to understanding the phenomena of somatization using the knowledge of medicine and psychology to treat human being. A Brief Group Psychanalytic Psychotherapy (BGPP) for psychosomatic patients has been used to supplement the treatment of some diseases including Systemic Lupus Erythematosus (SLE). The hypothesis of the study is that BGPP beside clinical treatment can improve the quality of life and coping in SLE patients. The aim of the study is to evaluate the effectiveness of BGPP in Brazilian SLE patients.

Primary objective: To evaluate the effectiveness of BGPP to improve quality of life. Secondary objectives: To evaluate the effectiveness of BGPP to improve coping, anxiety and depression symptoms. SLE patients will be randomized to receive Psychotherapy or only clinical treatment. The effectiveness will be assessed through specific questionnaires.

DETAILED DESCRIPTION:
This is a prospective randomized clinical trial. Patients with SLE (ACR criteria, 1997) treated at Rheumatology Division out-patient clinic of a university hospital were enrolled. A sample of 80 patients was assessed at the beginning of the study (baseline) and will be re-evaluated after 20 weeks (final) by clinical and psychological scales. Patients were randomized by computer program and divided into experimental group (EG) and control group (CG). Patients of both groups continued their medical treatment at the clinic. EG will be treated with BGPP for 20 sessions once a week for 20 consecutive weeks in small groups. The control group will be on a waiting list until the end of the study and will be treated subsequently.

Inclusion criteria:

* Female gender
* Four or more ACR criteria for classification of SLE
* Age above 18 years
* Follow-up at the clinic for at least 6 months

Exclusion criteria :

* Illiterate patients
* Mental or physical comorbidities that compromise their participation

Evaluation:

The following scales (adapted and validated for Portuguese Language) were being applied for a blinded evaluator to assess patients at baseline and after 20 weeks:

* Systemic Lupus International Disease Activity - SLEDAI Bombardier,1992);
* Systemic Symptom Checklist (SSC)(Freire, 2008);
* Systemic Lupus Erythematosus Quality of Life - SLEQOL (Freire, 2008);
* Coping strategies inventory of Folkman and Lazarus (Savoia,1996).
* Hospital Anxiety and Depression (Botega, 1995);
* Vital events scale of Holmes and Rahe (1967) (Savoia, 1995) and

Comparisons inter and intra groups were being analyzed using the Q square test for categorical variables and Student's t test, Mann-Whitney, Wilcoxon or ANOVA for quantitative variables. P values <0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Female patients,
* SLE (ACR criteria)
* over 18 years old
* followed up at the clinic for at least 6 months

Exclusion Criteria:

* illiterate patients,
* patients with mental or physical comorbidities that compromise their participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 20 weeks
  Significant improvement of scores of SLEQOL questionnaire

SECONDARY OUTCOMES:
Coping | 20 weeks
  Coping were assessed by Coping strategies inventory of Folkman and Lazarus.

OTHER OUTCOMES:
anxiety and depression | 20 weeks
  these variables will be assessed by Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Emilia I Sato, MD, PhD, Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Conceicao CTM, Meinao IM, Bombana JA, Sato EI. Psychoanalytic psychotherapy improves quality of life, depression, anxiety and coping in patients with systemic lupus erythematosus: a controlled randomized clinical trial. Adv Rheumatol. 2019 Jan 22;59(1):4. doi: 10.1186/s42358-019-0047-y. PMID 30670099